CLINICAL TRIAL: NCT01776021
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Trial to Assess the Effects of a Cranberry Beverage on Women With Recent History of Urinary Tract Infections
Brief Title: Effects of a Cranberry Beverage on Women With Recent History of Urinary Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ocean Spray Cranberries, Inc. (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRV-1201
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2013-11

CONDITIONS: Urinary Tract Infections; Infection; Urologic Diseases
Keywords: Urinary tract infection; Recurrent urinary tract infection; Cranberry; Prevention; E-coli
MeSH Terms: conditions — Urinary Tract Infections; Infections; Urologic Diseases; Escherichia coli Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cranberry juice (Active Comparator): cranberry juice beverage at a dose of one 8 oz. beverage per day for six months
  Interventions: Other: cranberry juice
- Placebo (Placebo Comparator): placebo beverage at a dose of one 8 oz. beverage per day for six months
  Interventions: Other: placebo beverage

INTERVENTIONS:
Other: cranberry juice — cranberry juice beverage at a dose of one 8 oz. beverage per day for six months
  Arms: cranberry juice
Other: placebo beverage — placebo beverage at a dose of one 8 oz. beverage per day for six months
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects of a cranberry juice beverage on rates of Urinary tract infection (UTI) recurrence in women with a history of UTI.

DETAILED DESCRIPTION:
Urinary tract infections (UTI) are the second most common infection of any organ system and the most common urological disease in the United States, with a total annual cost of more than $3.5 billion. Although UTIs can occur in both men and women, they are about 50 times more common in adult women than adult men. It is estimated that 25% of women diagnosed with a primary UTI will suffer a recurrence within two to three months. While no universal definition has been accepted, recurrent UTI is usually defined as three episodes in the last 12 months or two episodes in the last six months following initial infection. In an estimated 75 to 95% of cases of uncomplicated UTI, Escherichia coli (E. coli) is the underlying cause.

Cranberries have historically been associated with urinary tract health, but only recently has the biologic plausibility of cranberry use in the prevention of UTI been addressed. Current research suggests that A-type proanthocyanidins, a specific class of polyphenolic compounds found uniquely abundant in cranberries, inhibit adhesion of bacteria (including multidrug resistant E.coli) to cultured epithelial cells of the urinary tract.

This study will compare the effects of a cranberry juice beverage vs placebo on rates of UTI recurrence in women with a history of UTI.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has had at least 2 episodes of a UTI treated by a healthcare professional in the last year and at least 1 treated UTI within the last 6 months.
2. Subject is willing to avoid listed Vaccinium products (including cranberry juice, cranberries, craisins, blueberries, cranberry/blueberry powders, pills, or supplements, probiotics) for 2 weeks prior to enrollment and throughout intervention.
3. Subject agrees to avoid probiotic dietary supplements for 2 weeks prior to enrollment and throughout intervention.
4. Subject agrees to limit all probiotic-containing foods/yogurt and yogurt-containing products to no more than an 8 oz serving/d within 2 weeks prior to enrollment and throughout intervention.
5. Subject is willing to limit all soda, pop or energy drinks (diet or regular sweetened) to < 20 oz/d within 2 weeks prior to and throughout intervention.

Exclusion Criteria:

1. Subject has an in-dwelling catheter, polycystic disease, interstitial cystitis, previous urological surgery, stones, or anatomical abnormalities of the urinary tract, spinal cord injury, immuno-compromised conditions, severe renal impairment, or multiple sclerosis.
2. Subject has a history of antibiotic prophylaxis use for UTI. A 2-week washout period prior to enrollment will be allowed.
3. Subject has a body mass index (BMI) >40.0 kg/m2.
4. Subjects with diabetes mellitus and HbA1C >8.0% prior to enrollment.
5. Subject has diabetes mellitus treated with insulin.
6. Subject has an active infection or sign/symptoms of an infection (i.e., including a UTI).
7. Subject has used oral anti-coagulants within the last 4 weeks.
8. Subject has a history or presence of cancer in the prior two years, except for nonmelanoma skin cancer.
9. Subject is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable will be UTI incidence density, defined as the semi-annualized number of UTIs in each group, adjusted for susceptible time under observation. | six months

SECONDARY OUTCOMES:
Time from randomization to first clinical UTI. Time from randomization to first clinical UTI w/ pyuria. Time from randomization to first clinical UTI w/ microbiological verification. The fraction of subjects w/ one or more episode(s) of clinical UTI. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — Biofortis Clinical Research, Inc.
Locations (17):
- United States (17):
  - Chandler, Arizona
  - Scottsdale, Arizona
  - San Diego, California
  - Santa Rosa, California
  - Denver, Colorado
  - Edgewater, Florida
  - Miami, Florida
  - Summerfield, Florida
  - Ocean Spray Cranberries Research Sites, Addison, Illinois
  - Evanston, Illinois
  - Edina, Minnesota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Anderson, South Carolina
  - Dallas, Texas
  - Pleasant Grove, Utah
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952
- [Derived] Straub TJ, Chou WC, Manson AL, Schreiber HL 4th, Walker BJ, Desjardins CA, Chapman SB, Kaspar KL, Kahsai OJ, Traylor E, Dodson KW, Hullar MAJ, Hultgren SJ, Khoo C, Earl AM. Limited effects of long-term daily cranberry consumption on the gut microbiome in a placebo-controlled study of women with recurrent urinary tract infections. BMC Microbiol. 2021 Feb 18;21(1):53. doi: 10.1186/s12866-021-02106-4. PMID 33596852
- [Derived] Maki KC, Kaspar KL, Khoo C, Derrig LH, Schild AL, Gupta K. Consumption of a cranberry juice beverage lowered the number of clinical urinary tract infection episodes in women with a recent history of urinary tract infection. Am J Clin Nutr. 2016 Jun;103(6):1434-42. doi: 10.3945/ajcn.116.130542. PMID 27251185